CLINICAL TRIAL: NCT06922968
Title: Standard Versus Transrectal Ultrasound (TRUS)-Guided Endoscopic Treatment of Benign Prostatic Hyperplasia: A Prospective Randomized Controlled Trial
Brief Title: Real-Time (TRUS) Guidance in Endoscopic Treatment of BPH
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohamed ElSharkawy, Principal Investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TRUS with TURP and enucleation
Record Dates: First submitted 2025-03-17; First posted 2025-04-11 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2025-04

CONDITIONS: BPH (Benign Prostatic Hyperplasia)
MeSH Terms: conditions — Prostatic Hyperplasia

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Experimental): Control cases under went TURP and enucleation
  Interventions: Procedure: Standard TURP and enucleation
- TRUS Guided group (Experimental): TRUS guided group during TURP and enucleation
  Interventions: Procedure: TRUS-Guided TURP and enucleation

INTERVENTIONS:
Procedure: TRUS-Guided TURP and enucleation — realtime TRUS guidance during the procedure (TURP and enucleation)
  Arms: TRUS Guided group
Procedure: Standard TURP and enucleation — No TRUS guidance during the procedure (TURP and enucleation)
  Arms: Control group

SUMMARY:
The study aims to evaluate the role of TRUS in improving the efficacy and safety of endoscopic enucleation of prostate and TURP.

DETAILED DESCRIPTION:
Standard TURP is an established procedure for managing BPH but has limitations, including the risk of incomplete adenoma removal and complications such as bleeding. Research on transurethral enucleation techniques has demonstrated potential for improved outcomes, especially in larger prostates. However, challenges persist in achieving precise resection boundaries and minimizing intraoperative risks.

TRUS, widely utilized for prostate biopsy and volume assessment, has recently gained attention for its intraoperative applications. Studies show that real-time TRUS provides accurate imaging of prostate anatomy and resection planes, helping surgeons better differentiate adenomatous tissue from surrounding structures. This enhances surgical precision, reduces intraoperative bleeding, and minimizes residual tissue, leading to better outcomes in procedures like TURP and enucleation.

Current TURP and enucleation approaches depend heavily on endoscopic visual guidance, which, despite significant advancements, can lead to residual tissue, excessive bleeding, and prolonged recovery. While enucleation techniques have addressed some of these challenges, they remain less accessible due to high costs and steep learning curves, making them unsuitable for all healthcare settings.

Integrating TRUS into TURP or enucleation offers the potential to address these limitations by enhancing tissue differentiation and guiding precise resection. This study aims to evaluate the efficacy of TRUS in reducing complications, achieving complete tissue removal, and improving patient recovery outcomes, potentially paving the way for its routine adoption in BPH surgery.

ELIGIBILITY:
Inclusion Criteria:

* Male patients aged 50-80 years
* Diagnosed with benign prostatic hyperplasia (BPH) and scheduled for TURP or prostatic adenoma enucleation.
* The patients have clear indication for endoscopic surgery (according to the guidelines).
* Clinically fit patients for surgery.
* Signed an informed consent.

Exclusion Criteria:

* • Prostate cancer

  * Previous urethral or prostate surgery
  * Neurogenic bladder
  * Urethral stricture

Ages: 50 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 114 (Estimated)
Dates: Start 2025-04-01 (Estimated); Primary Completion 2026-10-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
efficacy of endoscopic treatment of BPH | At 12 weeks after the procedure
  Intervention efficacy will be evaluated by comparing the Peak flow rate in ml/second.(measured by uroflowmetry) between the two groups

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Mohamed Abdel-Moniem Hassanein, professor of Urology, Study Director — Assiut University
Locations (1):
- Assiut university, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No
to put protect privacy of participants